CLINICAL TRIAL: NCT06450691
Title: Modeling of Amyotrophic Lateral Sclerosis Using Patient Fibroblasts to Study Different Form of the Disease.
Brief Title: Modeling Amyotrophic Lateral Sclerosis With Fibroblasts
Acronym: FIBRALS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP231795
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; genetic; fibroblasts
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (SLA, healthy controls and asymptomatics) (Experimental): Patients fulfilling the El Escorial criteria definite ALS or asymptomatics or Healthy controls
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — skin biopsy and blood sampling

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is the most common motor neuron disease in adults. This longitudinal study involves three cohorts of participants: patients with sporadic or hereditary ALS, asymptomatic individuals carrying pathogenic mutations responsible for ALS, and control subjects. In this study, a skin biopsy and blood sampling will be performed at the initial visit (M0), then at M12 (+/- 2 months) for patients, and at M36 (+/- 12 months) for asymptomatic carriers of pathogenic mutations. The aim of this research is to model ALS pathology using fibroblasts derived from the patients' skin biopsies.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is the most common motor neuron disease in adults. This longitudinal study involves three cohorts of participants: patients with sporadic or hereditary ALS, asymptomatic individuals carrying pathogenic mutations responsible for ALS, and control subjects. In this study, a skin biopsy and blood sampling will be performed at the initial visit (M0), then at M12 (+/- 2 months) for patients, and at M36 (+/- 12 months) for asymptomatic carriers of pathogenic mutations. The aim of this research is to model ALS pathology using fibroblasts derived from the patients' skin biopsies.

ELIGIBILITY:
Inclusion criteria common to all 3 populations:

* adults, both sexes
* with written consent to participate in the study
* affiliated to a social security scheme

ALS patients :

* patients with ALS according to the revised El Escorial criteria :
* with a hereditary form of ALS, defined by the presence of a family history of ALS or by the demonstration of a pathogenic mutation in the patient or
* with a juvenile form of the disease, defined by onset of symptoms at less than 30 years of age or
* with a sporadic form of ALS

Asymptomatic mutation carriers :

- Asymptomatic individuals who carry a mutation causing ALS but have not developed symptoms.

Healthy subjects:

* control individuals, taking into account male/female and close age matching

Exclusion Criteria:

* with a known skin disease (acne, atopic dermatitis, psoriasis, melanoma, skin carcinoma, rosacea, scabies; as referenced on http://dermato-info.fr/), which in the investigator's opinion constitutes a contraindication to skin biopsy
* have a platelet count of less than 75,000/mm3 in a laboratory test less than 3 months old,
* with a proven allergy to lidocaine or prilocaine,
* Pregnant or breast-feeding women, or subjects under guardianship, curatorship or safeguard of justice.
* Patient's condition which, in the opinion of the investigator, is incompatible with skin sampling or participation in the study.
* Participation in a clinical trial (involving a drug) or other interventional research if this interferes with FIBRALS research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2033-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Detection of cytoplasmic TDP-43, TIA1 and/or p62 aggregates in patient fibroblasts | 1 year
  Detection of cytoplasmic TDP-43, TIA1 and/or p62 aggregates in patient fibroblasts subjected to various cellular stresses by immunofluorescence analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Neurosciences, Paris, France